CLINICAL TRIAL: NCT02455830
Title: A Study to Determine if Autologous Umbilical Cord Blood Cell Therapy Alters Serum Levels of Cytokines and Trophic Factors in Neonatal Encephalopathy
Brief Title: Cytokines Associated With Cord Blood Cell Therapy for Neonatal Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Neonatal Encephalopathy Consortium, Japan (Network)
Collaborators: Osaka City University (Other); Yodogawa Christian Hospital (Other); Kurashiki Central Hospital (Other); Nagoya University (Other); Osaka City General Hospital (Other); Saitama Medical University (Other); National Cerebral and Cardiovascular Center, Japan (Other); National Center for Child Health and Development, Japan (Unknown); Tokyo University (Other); Tokyo Women's Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: UMIN000014903-Cytokines
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Neonatal Encephalopathy (Neonatal Hypoxic-ischemic Encephalopathy)
Keywords: Neonatal encephalopathy; Hypoxic-ischemic encephalopathy; Newborn infants; Cytokines; Trophic factors
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cell-treated: Infants with encephalopathy who receive autologous umbilical cord blood cell therapy along with therapeutic hypothermia.
  Interventions: Biological: Autologous cord blood cell therapy
- Cooled only: Infants with encephalopathy who receive therapeutic hypothermia only.

INTERVENTIONS:
Biological: Autologous cord blood cell therapy — The neonates receive their own non-cryopreserved volume- and red blood cell-reduced cord blood cells. The cord blood cells are divided into 3 doses and intravenously infused at 12-24, 36-48, and 60-72 hours after the birth.
  Groups: Cell-treated

SUMMARY:
This is a observational study to assess the effects of and to explore the mechanisms of autologous umbilical cord blood cell therapy for neonatal encephalopathy by way of measuring serum cytokines.

DETAILED DESCRIPTION:
The effects and mechanisms of umbilical cord blood cell therapy for perinatal brain injury are not well understood. This is a multicenter study to measure serum levels of inflammatory cytokines and trophic factors associated with perinatal brain injury and repair in term gestation newborns with neonatal encephalopathy (hypoxic-ischemic encephalopathy). This study proceeds along with the study "Autologous cord blood cell therapy for neonatal encephalopathy (ClinicalTrials.gov identifier: NCT02256618)". Blood samples are obtained before the first cell infusion, and subsequently 2h, 24h, 48h, and 7 days after the first cell infusion. Blood samples are obtained in the same manner from newborns with neonatal encephalopathy who are not receiving the cell therapy.

ELIGIBILITY:
Inclusion Criteria:

Infants are eligible if they meet all the following inclusion criteria except 4.

1. ≥36 weeks gestation
2. Either a 10-minute Apgar score ≤5, continued need for resuscitation for at least 10 minutes, or severe acidosis, defined as pH <7.0 or base deficit ≥16 mmol/L in a sample of umbilical cord blood or any blood during the first hour after birth
3. Moderate to severe encephalopathy (Sarnat II to III)
4. A moderately or severely abnormal background amplitude-integrated EEG (aEEG) voltage, or seizures identified by aEEG, if monitored
5. Up to 24 hours of age
6. A person with parental authority must have consented for the study.

Exclusion Criteria:

1. Known major congenital anomalies, such as chromosomal anomalies, heart diseases
2. Major intracranial hemorrhage identified by brain ultrasonography or computed tomography
3. Severe growth restriction, with birth-weight less than 1800 g
4. Severe infectious disease, such as sepsis
5. Infants judged critically ill and unlikely to benefit from neonatal intensive care including hypothermia by the attending neonatologist

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with encephalopathy who meet the inclusion criteria of therapeutic hypothermia, either those who receive the cell therapy or those who do not.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Changes in serum levels of cytokines and trophic factors | From birth up to 10 days of age

SECONDARY OUTCOMES:
Association with neuroimaging and neurodevelopmental functional outcome | 18 months
  Neuroimaging at 12 months of age and neurodevelopmental function at 18 months of age will be assessed whether they are associated with serum levels of cytokines and trophic factors during the early neonatal period.

CONTACTS AND LOCATIONS:
Overall Officials: Haruo Shintaku, MD, PhD, Study Director — Osaka City University Graduate School of Medicine
Locations (6):
- Japan (6):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Saitama Medical Center, Kawagoe, Saitama
  - Yodogawa Christian Hospital, Osaka
  - Osaka City General Hospital, Osaka
  - Osaka City University Hospital, Osaka